CLINICAL TRIAL: NCT00267527
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind, Phase 2 Study to Evaluate the Efficacy and Safety of CJC 1295 Administered for 12 Weeks in HIV Infected Patients With HIV Associated Visceral Obesity
Brief Title: A Study to Evaluate CJC 1295 in HIV Patients With Visceral Obesity
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: ConjuChem (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GH100-013
Record Dates: First submitted 2005-12-20; First posted 2005-12-21 (Estimated); Last update posted 2006-10-16 (Estimated); Status verified 2006-10

CONDITIONS: Obesity; HIV Infections
Keywords: Treatment Experienced; HIV Visceral Obesity
MeSH Terms: conditions — Obesity; HIV Infections | interventions — CJC 1295

INTERVENTIONS:
Drug: CJC 1295

SUMMARY:
This is a multicenter, randomized, placebo-controlled, double-blind, Phase 2 study. Patients will be treated for a total of 12 weeks. There will be a 6 week follow-up period after the treatment period ends. Patients will be randomly assigned to low dose CJC 1295, high dose CJC 1295 or placebo.

The objective is to assess and compare the efficacy, pharmacokinetics, safety, and tolerability of CJC 1295 in patients with human immunodeficiency virus (HIV) associated visceral obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 on stable antiviral regimen
* Documented HIV infection
* HIV associated visceral obesity
* Body mass index (BMI) > 24 and < 30 kg/m2

Exclusion Criteria:

* Diabetes
* Use of growth hormone (GH) or other GH secretagogues
* Use of systemic glucocorticoids,
* Use of megestrol acetate or other appetite stimulants,
* Use of general anorexigenic or weight-reducing agents, or
* Use of androgens, other than testosterone replacement therapy for male hypogonadism at physiological doses and on a stable regimen for at least 6 months prior to randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-12; Study Completion 2006-09